CLINICAL TRIAL: NCT05619692
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of SAGE-718 in Participants With Mild Cognitive Impairment or Mild Dementia Due to Alzheimer's Disease
Brief Title: A Study to Evaluate the Effects of SAGE-718 in Participants With Mild Cognitive Impairment or Mild Dementia Due to Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 718-CNA-202
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Alzheimer's Disease
Keywords: SAGE-718; Cognitive dysfunction; N-methyl-D-aspartate (NMDA)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAGE-718 (Experimental): Participants will receive SAGE-718, 1.2 milligrams (mg), orally, once daily (QD) for the first 6 weeks (Days 1 to 42), followed by 0.9 mg of SAGE-718 for the remainder of the treatment period up to Day 84.
  Interventions: Drug: SAGE-718
- Placebo (Placebo Comparator): Participants will receive SAGE-718-matching placebo, orally, QD, throughout the treatment period up to Day 84.
  Interventions: Drug: SAGE-718-matching Placebo

INTERVENTIONS:
Drug: SAGE-718 — Softgel lipid capsules.
  Arms: SAGE-718
Drug: SAGE-718-matching Placebo — Softgel lipid capsules.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the effect of SAGE-718 on cognitive performance in participants with Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the following criteria for mild cognitive impairment (MCI) or mild dementia due to Alzheimer's Disease (AD) at Screening:

   1. A memory complaint reported by the participant or their study partner
   2. A Clinical Dementia Rating (CDR) score of 0.5 to 1.0 (inclusive) with a memory box score ≥ 0.5
   3. Essentially preserved activities of daily living, in the opinion of the investigator
   4. Brain Magnetic Resonance Imaging (MRI) report, obtained within the 2 years preceding the Baseline Period, that is consistent with the diagnosis of AD with no clinically significant findings of non-AD pathology that could account for the observed cognitive impairment
2. Have a score of 15 to 25 (inclusive) on the Montreal Cognitive Assessment (MoCA) with years of education adjustment at Screening.

Exclusion Criteria:

1. Have participated in a previous clinical study of SAGE-718, have participated in a previous gene therapy study, or have received study treatment in any other drug, biologic, or device trial within 30 days or 5 half-lives (whichever is longer), unless the participant participated solely in the placebo arm of the study. Additionally, participants who have received treatment with antisense oligonucleotides (ASO) will be excluded
2. Have a condition that precludes undergoing an MRI, in accordance with standard operating procedures at the imaging facility (eg, ferromagnetic metal in the body, claustrophobia), in a participant requiring MRI during Screening
3. Have any medical or neurological condition (other than AD) that might be contributing to the participant's cognitive impairment or history of cognitive decline
4. Have a history, presence, and/or current evidence of

   1. Brain surgery, deep brain stimulation, or any history of hospitalization due to a brain injury
   2. Possible or probable cerebral amyloid angiopathy, according to the Boston Criteria
   3. Treatment with an anti-amyloid therapy (including biologics) without subsequent MRI demonstrating the absence of amyloid-related imaging abnormalities
   4. Seizures or epilepsy, with the exception of childhood febrile seizures
5. Participants has a history of suicidal behavior within 2 years or answers "YES" to Questions 3, 4, or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening or at Day 1 or is currently at risk of suicide in the opinion of the investigator
6. Have any of the following medical conditions:

   1. Any clinically significant finding on 12-lead electrocardiogram (ECG) during Screening in the opinion of the investigator
   2. Any clinically significant supine vital signs (heart rate, systolic and diastolic blood pressure) during Screening (note: vital sign measurements may be repeated once)
7. Have a history, presence, and/or current evidence of serologic positive results for human immunodeficiency virus (HIV)-1 or HIV-2, or hepatitis B or C
8. Have a positive pregnancy test, or be lactating, or intend to breastfeed during the study
9. Is known to be allergic to any of SAGE-718 excipients, including soy lecithin

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (37):
  - Sage Investigational Site, Gilbert, Arizona
  - Sage Investigational Site, Phoenix, Arizona
  - Sage Investigational Site, Lafayette, California
  - Sage Investigational Site, Long Beach, California
  - Sage Investigational Site, Redlands, California
  - Sage Investigational Site, San Diego, California
  - Sage Investigational Site, Sherman Oaks, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Hollywood, Florida
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Palm Beach Gardens, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Winter Park, Florida
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Savannah, Georgia
  - Sage Investigational Site, Honolulu, Hawaii
  - Sage Investigational Site, Meridian, Idaho
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Charlestown, Massachusetts
  - Sage Investigational Site, Methuen, Massachusetts
  - Sage Investigational Site, Chesterfield, Missouri
  - Sage Investigational Site, Papillion, Nebraska
  - Sage Investigational Site, Toms River, New Jersey
  - Sage Investigational Site, Albuquerque, New Mexico
  - Sage Investigational Site, Brooklyn, New York
  - Sage Investigational Site, Buffalo, New York
  - Sage Investigational Site, Staten Island, New York
  - Sage Investigational Site, Raleigh, North Carolina
  - Sage Investigational Site, Abington, Pennsylvania
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Nashville, Tennessee
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Dallas, Texas
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Fairfax, Virginia
- Puerto Rico (2):
  - Sage Investigational Site, Bayamón
  - Sage Investigational Site, Rio Piedras

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 40 investigative sites in the United States and Puerto Rico from 29 November 2022 to 09 July 2024.
Pre-assignment Details: 174 participants were randomized to receive either SAGE-718 or placebo, of which 4 participants were not treated.
Groups:
- Placebo: Participants received SAGE-718-matching placebo, orally, once daily (QD), throughout the treatment period up to Day 84.
- SAGE-718: Participants received SAGE-718, 1.2 milligrams (mg), orally, QD for the first 6 weeks (Days 1 to 42), followed by 0.9 mg of SAGE-718 for the remainder of the treatment period up to Day 84.
Period: Overall Study
Arm/Group | Placebo | SAGE-718
Started | 87 | 87
Completed | 79 | 77
Not Completed | 8 | 10
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Participant | 3 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Randomized but not treated | 1 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants in the Safety Set (which included all participants who were administered at least one dose of the investigational product [IP]) who had baseline and at least 1 post-baseline efficacy evaluation.
Groups:
- Placebo: Participants received SAGE-718-matching placebo, orally, QD, throughout the treatment period up to Day 84.
- SAGE-718: Participants received SAGE-718, 1.2 mg, orally, QD for the first 6 weeks (Days 1 to 42), followed by 0.9 mg of SAGE-718 for the remainder of the treatment period up to Day 84.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-718 | Total
Number analyzed (Participants) | 86 | 84 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (6.80) | 69.6 (6.83) | 69.6 (6.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 35 | 32 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 17 | 40
  Not Hispanic or Latino | 62 | 67 | 129
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 5 | 5 | 10
  Race: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Race: Black or African American | 14 | 6 | 20
  Race: White | 62 | 71 | 133
  Race: More than one race | 2 | 2 | 4
  Race: Unknown or Not Reported | 0 | 0 | 0
Wechsler Adult Intelligence Scale-IV (WAIS-IV) Coding Test Score [Mean (Standard Deviation); unit: score on a scale] — The WAIS-IV coding test is a valid and sensitive measure of cognitive dysfunction that correlates with real-world functional outcomes (e.g., the ability to accomplish everyday tasks) and recovery from functional disability, used to assess processing speed. The participant is required to identify the symbols matched to numbers using a key and write in the symbol beneath the associated number. The total score ranges from 0 to 135 and is based on the total number of codes correctly completed over a 120-second time limit. Higher scores indicate better processing speed. Population: Number analyzed is the number of participants with data available for analysis.
  score on a scale
    number analyzed (Participants) | 86 | 83 | 169
    (all) | 43.9 (14.44) | 46.5 (16.04) | 45.2 (15.26)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Wechsler Adult Intelligence Scale-IV (WAIS-IV) Coding Test Score
Description: The WAIS-IV coding test is a valid and sensitive measure of cognitive dysfunction that correlates with real-world functional outcomes (e.g., the ability to accomplish everyday tasks) and recovery from functional disability, used to assess processing speed. The participant is required to identify the symbols matched to numbers using a key and write in the symbol beneath the associated number. The total score ranges from 0 to 135 and is based on the total number of codes correctly completed over a 120-second time limit. Higher scores indicate better processing speed. Positive change from baseline indicates better processing speed. Least Squares (LS) Means were calculated using a mixed-effects model for repeated measures (MMRM) approach.
Time Frame: Baseline, Day 84
Population: FAS included all participants in the Safety Set (which included all participants who were administered at least one dose of the IP) who had baseline and at least 1 post-baseline efficacy evaluation. Overall number of participants analyzed indicates number of participants with data available for analysis at a specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 80 | 76
score on a scale | 3.8 (0.77) | 5.3 (0.79)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.1642, MRMM — The p-value was obtained using MMRM model which included treatment, visit, treatment-by-visit interaction as categorical covariates, and WAIS-IV at baseline as continuous covariates; Difference in LS Means = 1.5, 95% CI 2-sided [-0.64 to 3.73], Standard Error of Mean 1.11 — Difference was calculated as SAGE-718 - placebo

2. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as any AE on or after the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to Day 112
Population: The Safety Set included all participants who were administered at least one dose of the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 86 | 84
Participants | 50 | 42

3. Secondary Outcome: Number of Participants With at Least One TEAE by Severity
Description: A TEAE is defined as any AE on or after the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study. Severity was assessed as:
  * Mild: symptoms barely noticeable to participant or does not make participant uncomfortable; does not influence performance or functioning; prescription drug not ordinarily needed for relief of symptoms
  * Moderate: symptoms of a sufficient severity to make participant uncomfortable; performance of daily activity is influenced; participant is able to continue in study; treatment for symptoms may be needed
  * Severe: symptoms cause severe discomfort; symptoms cause incapacitation or significant impact on participant's daily life; severity may cause cessation of treatment with IP; treatment for symptoms may be given and/or participant hospitalized.
  Participant with multiple instances of events is counted only once using maximum intensity.
Time Frame: Up to Day 112
Population: The Safety Set included all participants who were administered at least one dose of the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 86 | 84
Participants
  Mild | 29 | 20
  Moderate | 19 | 20
  Severe | 2 | 2

4. Secondary Outcome: Number of Participants Who Withdrew From Study Due to TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as any AE on or after the first dose of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to Day 112
Population: The Safety Set included all participants who were administered at least one dose of the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 86 | 84
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to Day 112
Description: The Safety Set included all participants who were administered at least one dose of the IP.
Arm/Group | Placebo | SAGE-718
All-Cause Mortality (participants affected / at risk) | 1/86 | 0/84
Serious Adverse Events (participants affected / at risk) | 5/86 | 4/84
Other Adverse Events (participants affected / at risk) | 17/86 | 10/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=86) | SAGE-718 (N=84)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=86) | SAGE-718 (N=84)
Headache (Nervous system disorders) | 9 | 7
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dizziness (Nervous system disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT05619692/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT05619692/SAP_001.pdf